CLINICAL TRIAL: NCT01678365
Title: Safety and Efficacy of Single Daily Dose of Ceftriaxone and Metronidazole for Treatment of Complicated Appendicitis in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dan Miron, MD, Professor, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 043-07-EMC
Record Dates: First submitted 2012-07-24; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Complicated Appendicitis
Keywords: complicated appendicitis; Children; conservative therapy; Study population: Children 1 month - 14 years with Complicated appendicitis; Type of the study: prospective, open randomized
MeSH Terms: interventions — Ceftriaxone; Metronidazole; Ampicillin; Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ceftriaxone and metronidazole for complicated appendicitis. (Experimental): Children with complicated appendicitis treated with single daily dose of ceftriaxone and metronidazole.
  Interventions: Drug: ceftriaxone, metronidazole/ampicillin, gentamicin, and metronidazole
- Ampicillin, gentamicin, and metronidazole (Active Comparator): Children with complicated appendicitis treated with ampicillin, gentamicin, and metronidazole
  Interventions: Drug: ceftriaxone, metronidazole/ampicillin, gentamicin, and metronidazole

INTERVENTIONS:
Drug: ceftriaxone, metronidazole/ampicillin, gentamicin, and metronidazole

SUMMARY:
A prospective open randomized study conducted between July 1st 2008 and June 30th, 2009. Included were children younger than 14 years with Complicated appendicitis randomly assigned either to a single daily dose of Ceftriaxone and Metronidazole or Ampicillin, Gentamicin, and Metronidazole. The outcome variables compared were: maximum daily temperatures, overall duration of fever, time return to oral intake, length of antibiotic therapy, results of repeat WBC measure, general/intra abdominal complications, need for intra abdominal abscess drainage, Length of stay and adverse reaction.

DETAILED DESCRIPTION:
The study was conducted at the Pediatric Surgery Department at HaEmek Medical Center, Afula, Israel. Included were children age 1-14 years with complicated appendicitis that was defined by one of the followings: 1. Demonstration by abdominal ultrasound and/or computed tomography of appendix perforation and/or peri-appendicular abscess 2. Demonstration by abdominal ultrasound of free fluid, and signs of diffuse peritoneal irritation in the right lower quadrant of the abdomen 3. At surgery performed for suspected non complicated appendicitis. In a patient with perforate appendicitis that was diagnosed at surgery, appendectomy was performed by one of the 4 senior pediatric surgeons on call at the time of the child's admission. Exclusion criteria were: documented allergy to any of the study medications, acute or renal insufficiency at admission, and severe septic shock at admission.

Therapeutic approach: After the diagnosis of complicated appendicitis was established, patients were randomly assigned to therapy with either once daily of ceftriaxone and metronidazole or ampicillin, gentamicin and metronidazole. Therapy was change to piperacillin/tazobactam in patients who were still febrile at day 7-10 of the admission (if not given before), based on the clinical situation, and in all febrile patients at 11 day of the admission . All patients had also been treats after inclusion with pain control medications, no oral food or fluid , and intravenous hydration as necessary. Nasogastric tubes were not used routinely. On the fifth admission day patients who were stable, a febrile, could tolerate diet and had Complete blood count within normal limits were discharged home with oral amoxicillin/clavulanate therapy for further 7 days.

Follow-up at the admission: CBC and renal and liver function tests were obtained before starting the antibiotic treatment and repeated on day 4 in all patients. In the group treated with AGM, serum trough gentamicin concentration was drawn before the fourth dose with normal level considered as < 2 mcg/ml. Other blood studies were performed based on the discretion of the attending physician based on the patient's clinical status. For patients who were either febrile or had leukocytosis, at day 5 of therapy abdominal ultrasound was obtained to assess for the presence of an abscess. Patients in whom abscesses were delectated undergone per coetaneous drainage (when possible). The original antibiotic regimen was either continued or changed to piperacillin/tazobactam based on the clinical situation. Patients, in whom appendectomy had not been done at admission, were readmitted for appendectomy at 6 weeks. All patients had been followed for a year since the admission for signs of intra abdominal complication such: repeat abscess formation, repeat admission, obstruction etc.

Data collection: Data were recorded were: patient's age, weight, gender, maximum daily temperature, duration of fever, results of complete blood count, renal and liver function tests, gentamicin levels (where applicable), intra abdominal complications and duration of hospitalization. The outcome variables included maximum daily temperatures for each of the first 10 postoperative days, time to initial oral intake, length of hospitalization, length of antibiotic therapy, abscess formation rate, need to change antibiotic regimen, wound infection rate, and any abnormal findings during the follow-up visits.

Statistical analysis: Since data in the literature show that there is no difference of the length of stay in between the 2 regimens (in children with complicated appendicitis following operation), and most studies included relatively low number of patients, no power analysis was calculated. The difference between various parameters in the two treatment groups were assessed by 2 independent sample T tests or Fisher exact tests for categorical data and 2 independent sample t test or the Mann Whitney test for continuous data. Descriptive statistics were calculated as mean ± SD.

ELIGIBILITY:
Inclusion Criteria:

* Children age 1-14 years CA that was defined by one of the followings:

  1. Demonstration by abdominal ultrasound (US) and/or computed tomography (CT) of appendix perforation and/or peri-appendicular abscess
  2. Demonstration by abdominal ultrasound (US) of free fluid, and signs of diffuse peritoneal irritation in the right lower quadrant of the abdomen 3

Exclusion Criteria:

* Documented allergy to any of the study medications, acute or renal insufficiency at admission, and severe septic shock at admission.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Length of stay (days) | From admission to discharge from of first admission (if there are more than one), an expected average 2 weeks
Change of primary antibiotic regimen to Piperacillin/tazobactam | From admission to discharge from of first admission (if there are more than one), an expected average 2 weeks

SECONDARY OUTCOMES:
Number of new intrabdominal abcesses | From admission to discharge from of first admission (if there are more than one), an expected average 2 weeks

OTHER OUTCOMES:
Re hospitalization due to intra abdominal abcess formation | Within 2 years after day of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Surgery Department, HaEmek Medical Center, Afula, Israel